CLINICAL TRIAL: NCT02070666
Title: Preventive Strategies in Acute Respiratory Distress Syndrome
Brief Title: Preventive Strategies in Acute Respiratory Distress Syndrome (ARDS)
Acronym: EPALI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment and published data with no benefit
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Antonio Artigas Raventós, Director of Critical Care Arrea, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPALI
Record Dates: First submitted 2014-02-19; First posted 2014-02-25 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: ARDS
Keywords: ARDS; Prevention; Protective mechanical ventilation; low tidal volumes
MeSH Terms: interventions — Control Groups; Respiratory Dead Space

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Protective ventilation arm (Experimental): * Low tidal volumes (from 4 to 6 milliliters(mL)/kilogram (kg) of predicted body weight (PBW)
  * Plateau pressure less than 25 centimeter of water (cmH2O)
  * Minimum PEEP of 5 cmH2O.
  Interventions: Behavioral: Protective mechanical ventilation; Other: Dead space
- Control group (Active Comparator): Traditional-sized tidal volumes (from 8 to 10 mL/kg PBW)
  * Plateau pressure less than 25 cmH2O
  * Minimum PEEP of 5 cmH2O.
  Interventions: Behavioral: Control group; Other: Dead space

INTERVENTIONS:
Behavioral: Protective mechanical ventilation — Ventilation mode: volume control, pressure control, dual modes (It is allowed to change to a spontaneous mode; a minimum of 5 cmH2O level of support should be used; in case the resulting tidal volume exceeds 6 mL/kg PBW this is accepted. This is not a reason to use more sedation and/or muscle relaxants, or to switch the ventilator to a controlled mode of ventilation).
  * Tidal volume: 6 mL/Kg PBW, decreasing 1 mL/kg PBW each step if necessary (steps of 5 minutes), to maintain plateau pressure < 25 cmH2O until a minimum tidal volume of 4 mL/Kg PBW, unless the patient suffers from severe dyspnea or unacceptable acidosis.
  * Fraction of inspired oxygen inspired oxygen fraction (FiO2) > 0.21 to maintain oxygen saturation 90-92%.
  * PEEP ≥ 5 cmH2O, and optimized to maintain Oxygen saturation (SpO2) 90-92% (left to the discretion of the attending physician).
  * Plateau pressure ≤ 25 cmH2O
  Arms: Protective ventilation arm
Behavioral: Control group — Ventilation mode: volume control, pressure control, dual modes (It is allowed to change to a spontaneous mode, with the level of support adjusted to reach tidal volumes minimum of 8 mL/kg predicted body weight PBW; if it is not possible, the data collection should be continue and an intention-to-treat analysis will be done).
  * Tidal volume: minimum 8 mL/kg PBW. It is possible to increase until 10 mL/kg PBW unless plateau pressure increases above 25 cmH2O.
    · FiO2 > 0.21 to maintain oxygen saturation 90-92%.
  * PEEP ≥ 5 cmH2O, and optimized to maintain SpO2 90-92% (left to the discretion of the attending physician).
  * Plateau pressure ≤ 25 cm H2O.
  Arms: Control group
Other: Dead space — Volumetric capnography will be used. Dead space (Vd/Vt) measurements will be taken at baseline and daily after initiation of mechanical ventilation. Nursing and respiratory care activities (including changes to ventilator settings) will be suspended for at least 5 minutes prior to all Vd/Vt measurements.

SUMMARY:
The investigators hypothesis is that patients at risk of ARDS, detected by LIPS (Lung Injury Prediction Score), under mechanical ventilation could benefit from a protective ventilatory strategy (used in ARDS treatment) in order to avoid or decrease the ARDS development. This would lead to a decrease in incidence, mortality and health care costs associated to this syndrome.

This study will help to confirm the current evidence about low tidal volumes, evaluating adverse events of this strategy.

DETAILED DESCRIPTION:
The main objective is to evaluate the effect of a protective ventilatory strategy by using lower tidal volumes compared to the use of traditionally volumes in ARDS development.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 12 hours after start of invasive mechanical ventilation (MV) and admitted to participating ICU (it is recommended an inclusion as soon as possible during the first 3 hours).
* LIPS > 4 points.
* Absence of mild, moderate and severe ARDS criteria (Berlin definition).
* Older than 18 year-old.
* Signed informed consent

Exclusion Criteria:

* Bilateral pulmonary infiltrates in chest X-ray at admission.
* Mechanical ventilation > 12 hours.
* Previous pneumonectomy or lobectomy.
* Severe cranial trauma (Glasgow Coma Scale<9) or cranial hypertension.
* Severe chronic pulmonary disease (GOLD IV).
* Admission from other hospital under MV.
* Limitation of therapeutic effort.
* Pregnancy.
* Acute pulmonary embolism.
* Participation in other interventional trials.
* Previous randomized in the proposed trial.
* Absence of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-05; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
ARDS development | 7 days
  To determine the effect of a protective mechanical ventilation strategy using lower tidal volumes as compared to mechanical ventilation using traditionally-sized tidal volumes on development of ARDS.

SECONDARY OUTCOMES:
Mortality | 90 days
  In-hospital mortality, 28-day mortality and 90-day mortality
Ventilator-free days | 28 days after admission
  From 1 to 28 days over 28 days in a month
Dead space | 7 days
  Volumetric capnography
Length of stay | participants will be followed for the duration of ICU (Intensive Care Unit) and hospital stay, an expected average of 4 weeks
  ICU stay and hospital stay
Pneumonia | 7 days
  Incidence of pneumonia
Atelectasis | 7 days
  Incidence of atelectasis

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Sabadell, CSUPT, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] de Haro C, Neto AS, Goma G, Gonzalez ME, Ortega A, Forteza C, Frutos-Vivar F, Garcia R, Simonis FD, Gordo-Vidal F, Suarez D, Schultz MJ, Artigas A. Effect of a low versus intermediate tidal volume strategy on pulmonary complications in patients at risk of acute respiratory distress syndrome-a randomized clinical trial. Front Med (Lausanne). 2023 Jun 7;10:1172434. doi: 10.3389/fmed.2023.1172434. eCollection 2023. PMID 37351068